CLINICAL TRIAL: NCT07032311
Title: Effect of Behavioral Intervention/Therapy to Reduce Diabetes and Liver Disease Risk Through Prescribed Digital Therapeutics Enabled by AI/ML Powered Predictive Analytics
Brief Title: Digital Behavioral Therapy to Reduce Diabetes and Liver Disease Risk
Acronym: SIPPA-QH_HHC-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SIPPA Solutions INC (Industry)
Collaborators: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIPPA-QH_HHC-2025-S1
Record Dates: First submitted 2025-06-19; First posted 2025-06-23 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; Prediabetes; Liver Disease
Keywords: Type 2 diabetes mellitus; Prediabetes; Digital therapeutics; Behavioral intervention; Smartphone app; GLP-1 receptor agonist; Fib-4 score; Randomized pilot trial; Metabolic dysfunction-associated steatotic liver disease (MASLD); Health navigator support; SIPPA Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Participants are randomized into four parallel groups in a 1:1:1:1 fashion, stratified by current GLP-1 receptor agonist use. Two groups receive standard diabetes care (with or without GLP-1 therapy), and two groups receive standard care plus the SIPPA Health app intervention (with or without GLP-1 therapy). All participants follow their assigned regimen concurrently over the 6-month study period.
Masking Description: This is an open-label trial; no participants, investigators, outcome assessors, or data analysts are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ARM 1: Control without behavioral treatment (No Intervention): ARM-1-G1: Patient subjects receiving standard care services without GLP-1 medication as part of the treatment regimen. ARM-1-G2: Patient subjects receiving standard care services with GLP-1 medication as part of the treatment regimen.
- AMR-2: Behavioral intervention (Experimental): ARM-2-G1: Patient subjects receiving standard care services without GLP-1 medication as part of the treatment regimen, and SIPPA Health behavioral intervention/therapy. ARM-2-G2: Patient subjects receiving standard care services that includes GLP-1 medication as part of the treatment regimen, and SIPPA Health behavioral intervention/therapy.
  Interventions: Device: Behavioral Treatment

INTERVENTIONS:
Device: Behavioral Treatment — Description: ARM-2-G1: Patient subjects receiving standard care services without GLP-1 medication as part of the treatment regimen, and SIPPA Health behavioral intervention/therapy. ARM-2-G2: Patient subjects receiving standard care services that includes GLP-1 medication as part of the treatment regimen, and SIPPA Health behavioral intervention/therapy.
  Arms: AMR-2: Behavioral intervention

SUMMARY:
This clinical trial aims to find out if a digital behavioral program, delivered through the SIPPA digital therapeutics app, can help improve blood sugar control and lower the risk of liver fibrosis in adults with type 2 diabetes who are at low to moderate risk for liver disease.

Main Research Question:

Can adding the SIPPA behavioral program to standard diabetes care lower HbA1c (a marker of blood sugar control) more than standard care alone?

Study Design:

The study has two groups (called "arms") for comparison:

Arm 1: Control Group Subgroup 1.1: Participants receiving standard care without GLP-1 medication. Subgroup 1.2: Participants receiving standard care with GLP-1 medication.

Arm 2: Intervention Group Subgroup 2.1: Participants receiving standard care without GLP-1 medication, plus the SIPPA behavioral program.

Subgroup 2.2: Participants receiving standard care with GLP-1 medication, plus the SIPPA behavioral program.

Researchers will compare outcomes across the matched groups in each arm to evaluate the impact of the SIPPA program.

What Participants Will Do:

All participants will have lab tests at the start of the study, at 3 months, and at 6 months. These tests include:

* HbA1c (a measure of average blood sugar levels),
* Fib-4 score (used to estimate liver fibrosis risk), and
* Liver enzyme tests.

Participants in the intervention group (Arm 2) will also:

* Use the SIPPA app daily to complete behavioral modules, track blood sugar
* levels, and log health behaviors (like diet and activity).
* Have weekly check-ins with a health navigator to support progress and stay on track with their diabetes treatment plan.

DETAILED DESCRIPTION:
Study Purpose and Objectives This study is designed to evaluate whether a smartphone-based behavioral intervention, called SIPPA Health, can enhance the effects of standard diabetes care-including for patients who are prescribed GLP-1 receptor agonists (a common injectable diabetes medication). SIPPA Health, guided by behavioral predictive analytics, delivers daily lifestyle coaching through an app, including exercise goals, meal logging, glucose tracking, and weekly remote check-ins with a trained health navigator.

The study will examine whether adding SIPPA to standard treatment improves blood sugar control, reduces liver fibrosis risk, supports weight management, and helps personalize diabetes care through digital tools. Specific objectives include:

Glycemic Control: Measure changes in hemoglobin A1c (HbA1c)-a long-term blood sugar marker between those who use the SIPPA app and those who receive standard care alone.

Liver Health: Measure Fibrosis-4 (Fib-4) index, an estimate of liver scarring, between those who use the SIPPA app and those who receive standard care alone.

Population-level Diabetes Risk Indicator: Assess whether there is a difference in the distributions between SIPPA users and patients receiving only standard care service; where the distribution will consider BMI change, A1c progression, glucose variability (time-in-range), and engagement with self-care activities.

AI Risk Stratification (Pilot): Test a machine learning model that classifies participants by clinical, behavioral, and social determinants of health data. The aim is to inform future personalized care plans.

Study Design

This is a randomized, controlled pilot trial lasting six months, involving 200 adult participants with either type 2 diabetes or prediabetes (defined as two consecutive HbA1c values between 5.8% and 6.5%). All participants receive standard diabetes care and are randomly assigned to one of two main groups:

ARM 1 (Control Group): Standard care alone. ARM 2 (Intervention Group): Standard care plus the SIPPA Health app.

Each group is further divided based on whether the participant is currently using a GLP-1 receptor agonist:

Subgroup G1: No GLP-1 therapy. Subgroup G2: On GLP-1 therapy.

This results in two study arms with four subgroups for the purpose of comparative study:

Control without GLP-1 (ARM 1-G1) Control with GLP-1 (ARM 1-G2) SIPPA without GLP-1 (ARM 2-G1) SIPPA with GLP-1 (ARM 2-G2)

All participants complete the same laboratory and survey assessments at baseline, 3 months, and 6 months. These include blood tests (A1c, liver enzymes, lipids), weight, and self-reported lifestyle data. SIPPA users also receive a smartphone app with daily reminders, educational content, and weekly coaching calls to support their self-care routines.

Outcome Measures Primary Clinical Outcome (6 Months) Change in HbA1c (%): The main measure of long-term blood glucose control.

Secondary Outcomes Fibrosis-4 (Fib-4) Index: A validated liver fibrosis score calculated from age, AST (aspartate aminotransferase), ALT (alanine aminotransferase), and platelet count.

Weight and Body Mass Index (BMI): Measured in pounds and kilograms per square meter.

Time-in-Range (%): The percentage of glucose readings within the healthy range (70-180 mg/dL), assessed by continuous glucose monitor (CGM) or glucose logbooks.

Composite Diabetes Risk Indicator (DRI): A novel index that integrates change in A1c, glucose variability, and adherence to self-care behaviors (e.g., step counts, app engagement). Participants are categorized into low, medium, or high risk for diabetes-related complications.

Exploratory Outcomes App Engagement: For SIPPA users, the study will track number of logins, modules completed, step counts, and minutes spent in coaching calls.

Subgroup Effectiveness: Analysis to identify which population groups (e.g., based on baseline self-efficacy or social factors) benefit most from SIPPA.

Safety and Tolerability: Adverse events, hypoglycemia, or any app-related issues will be monitored continuously. Data are reviewed by a safety board and institutional review body.

ELIGIBILITY:
Inclusion Criteria:

* English Proficiency with a Middle-school Reading Level
* Owning a smartphone or obtaining one on-loan basis during the study period, with a data plan and/or the ability to receive text messages
* Possess basic skills to operate an (Android) smartphone, if you want to receive behavior intervention/therapy in addition to the standard care service
* Willingness to Modify Behavior, Physical activity, and diet
* Age 22 to 65
* Diagnosed with diabetes and prediabetes with two or more blood work results since 2021 revealing alanine aminotransferase (ALT), aspartate aminotransferase (AST), and platelet count (ICD-10 code; Prediabetes: R73.03, Diabetes: E08-E13); whereas prediabetes is clinically defined as two consecutive measure of A1C between 5.8 and 6.5
* Willing to communicate with the project team via phone, email, or SMS once a week

Exclusion Criteria:

Consume more than one and a half times the limit of alcohol recommended for the population (15g/day for women and 30 g/day for men) (ICD-10 code: K70.9)

* Pregnancy (ICD-10 code: Z33.3)
* Receiving Hepatotoxic Medication (ICD-10 code: K76.1)
* Cirrhosis, Hepatitis B/C, and Other Chronic Liver Diseases (ICD-10 code: K.74, B19.10, B19.20, K72.1)
* Cardiovascular Events in the Past 6 Months and Symptomatic Heart Failure (ICD-10 code: I.21, I.25, I.50, I63.9)
* Stage 4 and Above Chronic Kidney Disease (CKD) and End-Stage Renal Disease (ESRD)(ICD-10 code: N18.4, N18.5, N18.6)
* Untreated Hypothyroidism (ICD-10 code: E03.9)
* Depression (ICD-10 code: F32.A)
* A patient who already received a digital behavioral intervention/therapy prescribed by a clinician is ineligible for this study for safety considerations.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline to 6 months after randomization
  Hemoglobin A1c is reported as a percentage (%) of glycosylated hemoglobin, with typical values ranging from approximately 4% (normal) up to >14% (poor control). Higher percentages indicate worse long-term glycemic control. Our primary outcome metric is the absolute difference in percentage points (e.g., a decrease from 8.1% at baseline to 7.2% at six months reflects a change of -0.9 percentage points).

CONTACTS AND LOCATIONS:
Locations (1):
- NYC Health + Hospitals/Queens Hospital Center Diabetes Center of Excellence, Jamaica, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sy B, Wassil M, Hassan A, Chen J. Personalizing self-management via behavioral predictive analytics with health education for improved self-efficacy. Patterns (N Y). 2022 May 17;3(6):100510. doi: 10.1016/j.patter.2022.100510. eCollection 2022 Jun 10. PMID 35755867